CLINICAL TRIAL: NCT00580281
Title: Effect of Imatinib on Bone Metabolism in Patients With Chronic Myelogenous Leukemia or Gastrointestinal Stromal Tumors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-142
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer; Leukemia; Chronic Myelogenous Leukemia
Keywords: Gastric cancer; Leukemia; Chronic Myelogenous Leukemia; Imatinib; Gleevec
MeSH Terms: conditions — Stomach Neoplasms; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- blood, urine, and dexa scan (Experimental): This study will involve venipuncture for obtaining blood samples; a spot second void (whenever possible) urine sample will be obtained at the same time. A Dexa scan to evaluate bone density will be obtained at the beginning, middle and end of the study.
  Interventions: Other: blood test, urine test, and bone density x-ray.

INTERVENTIONS:
Other: blood test, urine test, and bone density x-ray. — start of the study (month 0), and at months 3, 6, 9, 12 (1 year), 15, 18, 21, and 24 (2 years)

SUMMARY:
The drug that you are taking for your cancer, imatinib (GleevecTM), has recently been shown to have some new types of side effects. In some people, imatinib can affect how bones are made.

The purpose of this study is to find out if imatinib is causing these side effects in you. We can check how your bones form by testing your blood and urine. We can also check your bone strength by doing a special X-ray of your bone called bone density (or DEXA scan).

DETAILED DESCRIPTION:
Preliminary data from this institution suggest that imatinib, likely by inhibiting platelet derived growth factor receptor (PDGFR), inhibits bone formation and resorption in a high percentage of patients with either chronic myelogenous leukemia (CML) or gastrointestinal stromal tumors(GIST).1 Some, but not all, patients taking imatinib developed hypophosphatemia but the effect on bone, as measured by markers of bone synthesis and metabolism, was seen in some patients with normal phosphate levels as well. Marked urinary phosphate wasting with elevated levels of parathyroid hormone was seen in nearly all patients. The effect of imatinib on bone may be dose-related. Patients with hypophosphatemia were routinely started on oral phosphate replacement, but follow up determinations of urinary phosphate wasting were not performed.

The clinical consequences of these abnormalities on bone are not yet known. This trial will study 60 patients with CML in chronic phase, early accelerated phase (as detected by cytogenetics only) or GIST who are already taking imatinib. Parameters relating to bone metabolism will be checked every 3 months for 2 years. We will determine the incidence of bone abnormalities in this treated population, determine whether fasting serum phosphate can predict for changes in bone metabolism, determine whether there is change in bone density by measuring serial bone densitometry, determine whether oral phosphate replacement can restore phosphate balance, and determine whether there is a dose effect of imatinib on parameters of bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CML in chronic phase, accelerated phase based on cytogenetic abnormalities in addition to Philadelphia chromosome but with less than 5 % blasts, or GIST taking imatinib
* Patients with life expectancy of at least 12 months; patients must be on imatinib at time of study entry.
* Ability to sign informed consent and/or assent

Exclusion Criteria:

* Patients with a known parathyroid disorder; active thyroid disorder except stable, replaced hypothyroidism; Cushing's syndrome; uncontrolled diabetes mellitus (could have unexpected fluid, electrolyte and mineral shifts); sarcoidosis (elevated calcitriol levels from granulomata); hypercalcemia of malignancy (i.e., PTHrP-mediated or extensive bone mets);known tumor-induced osteomalacia; Paget's disease of bone; known X-linged or autosomal dominant hypophosphatemic rickets/osteomalacia; known renal tubular disease (e.g., Fanconi's syndrome); chronic GI malabsorption sydrome.
* Patients taking oral calcium in excess of calcium 750 mg and Vitamin D 400 mg daily (ie, that contained in a single multivitamin). Patients taking more than these amounts may be eligible for this study if vitamin and mineral supplementation in excess of this is stopped for a minimum of 2 weeks prior to study entry.
* Patients taking oral or intravenous steroids, calcitonin, any selective estrogen modulating agent such as tamoxifen or raloxifene, gallium nitrate, and other bone seeking radionuceotides, any calcimimetic agent such as cinacalet.
* Patients who have had prior treatment with cisplatin, carboplatin, oxaliplatin, ifosfamide, or cyclophosphamide.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
This pilot study will collect longitudinal data on bone metabolism for patients treated with imatinib. Sixty patients will be followed over a two-year period on this protocol, with bone marker assessments ascertained every 3 months (+2 weeks). | Every 3 months (+2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ellin Berman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org